CLINICAL TRIAL: NCT00163930
Title: Post-Operative Pain Management in Patients Undergoing Uterine Artery Embolisation for Symptomatic Leiomyomata
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Other Study IDs: AlfRad2004-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2005-09

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroids; embolisation; pain management
MeSH Terms: conditions — Leiomyoma; Agnosia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This project seeks to evaluate the effectiveness of a new post-operative pain relief program for women who have undergone uterine artery embolisation (UAE).

UAE is performed by an interventional radiologist as a treatment of uterine fibroids (non-cancerous growths of the uterus.) UAE can be associated with a high level of post-procedural pain and it is the purpose of this study to evaluate a new relief regimen for dealing with this acute pain.

There will be two treatment groups into which patients will be randomly assigned. One will receive the current post-operative therapy (dose-on-demand) and the other will receive the new therapy (pre-emptive dosing). Otherwise patients will receive standard management protocol for this procedure. Only patients that are scheduled for UAE will be enrolled (up to 40 patients).

The new treatment involves giving the patient their morphine dose orally and sixty minutes before the procedure begins (pre-emptive dosing) as opposed to current standard treatment which involves giving the patient a dose of morphine intravenously once they feel pain.

Information to be collected directly from patients includes pain and nausea levels, indicated on a visual scale (a 10 centimetre line showing a spectrum of no pain to worst pain imaginable) as well as their opinions of the effectiveness of the pain relief program and the procedure itself. This information is to be collected immediately post-procedure and at 2, 4, 6 and 24 hours post procedure. Each VAS will take the patient approximately 20 seconds to complete. Information about concurrent medication and procedure complications, post-operative vomiting and respiratory depression will be collected from the patient's history.

DETAILED DESCRIPTION:
Post operative Pain Management in Paitents Undergoing Uterine Artery Embolisation for Symptomatic Leiomyomata

Protocol (Ver 2.1)

1.1 Research Question Does pre emptive morphine dosing help reduce acute post operative pain (as expressed on a visual analogue scale, VAS) and/or post operative opioid use in patients undergoing uterine artery embolisation?

2.1 Enrolment Patients are enrolled by Prof Ken Thomson or Dr Stuart Lyon during a planning consultation with each woman. They will be required to sign a consent form if they choose to participate at this point. 3 photocopies of this consent form will be taken, with one copy to go with: the patient; the history; and the data file.

2.2 Exclusions

Patients with the following should be excluded from the study:

* Pregnancy
* Contrast allergy
* Allergy to one or more of the treatment drugs
* History of alcoholism
* Diagnosed hepatic disease
* Renal insufficiency
* Acute pelvic infection
* Endometrial carcinoma
* Undiagnosed pelvic mass
* Non English speaking patients
* Patients who require post op non opioid analgesia

3.1 Randomisation and blinding The placebo and oxycontinSR tablets have been pre randomised by the clinical trials pharmacy on LG level (Ann Mak).

4.1 Pre medications The trial drug (oxycontin) will be ordered on a yellow clinical trial prescription form. A day before the patient arrives, this form should be faxed to the Clinical Trials Pharmacy (Fax No 3305). A registered nurse from the ward or researcher should then pick up the drugs from the Clinical Trials Pharmacy on LG level.

The other non trial medications should be either already on the ward or should be ordered via pharmacy as per normal.

The trial drugs and pre medications will all be written up on a prepared drug chart which will be given to the ward.

4.2 Treatment

The ward staff will administer the drugs as prescribed on the drug chart 60 +/- 20 minutes prior to the procedure.

The differences in the treatment is shown on the following table. Dose on demand treatment Pre emptive treatment

1 hour before surgery:

* Paracetamol 1.5g
* Temazepam 20mg
* Placebo OxycontinSR
* Piroxicam (Feldene) 20mg
* Ondansetron 8mg 1 hour before surgery:
* Paracetamol 1.5g
* Temazepam 20mg
* OxycontinSR
* Piroxicam (Feldene) 20mg
* Ondansetron 8mg

Surgery:

* PCA morphine
* 1mg dose with 5 minute lockout Surgery:
* PCA morphine
* 1mg dose with 5 minute lockout Follow up
* Endone 5-10mg oral 4/24 prn Follow up
* Endone 5-10mg oral 4/24 prn

The ward staff will be blinded as to which treatment the patient receives since the pre meds are have been randomised and blinded by the pharmacy.

5.1 Post op Pain and nausea measurements will be taken at 2, 4, 6 and 24 hours using the visual analogue scale (VAS) questionnaire sheets. This can be done either by the researchers, or if time permits, ward staff.

Drug related side effects are also recorded, such as respiratory depression and vomiting and it is therefore important for these to be carefully documented in the patient's history.

5.2 Deviations from pain management protocol There may be instances where the PCA does not deliver adequate pain relief. It may be necessary in these cases to deviate from the pain management protocol for the comfort of the patient. This does not necessarily exclude the patient from the study. However, the way in which the data is interpreted once non opioid analgesia is given should be done with caution.

Deviations should be instituted when:

* Obvious drug related side effects are evident (e.g. respiratory depression, narcosis); or
* Pain is not at an acceptable level at 6 hours post procedure; or
* Pain is not at a level in keeping with routine post UAE pain as reported by nursing or medical staff.

Please notify Dr Stuart Lyon or Dr Jeff Tam (ex 3606) if the Pain Team needs to intervene for these patients. They will then assess whether or not the patient will be excluded from the study.

6.1 Discharge

When patients are deemed ready for discharge they need to take home a discharge pack with some questionnaires for them to fill out at home. These should be done at 24 hours post procedure. The pack will include:

* Pain VAS
* Nausea VAS
* Overall pain relief rating VAS
* UAE procedure rating VAS
* Instructions sheet
* Reply paid, self addressed envelope

Please check that the 2, 4 and 6 hour questionnaires have been filled out before the patient is discharged, and that they leave with the discharge pack. Once completed, the questionnaires should be sent back to the Radiology Research Department.

Most patients will be discharged within 24 hours of the procedure. In the event that the patient stays in hospital longer than 24 hours, then the discharge pack should be completed at the 24 hour mark. The completed data sheets should then be sent back to the Radiology Research Department.

If the data sheets are not received within 2 weeks of discharge, the researchers should make a phone call to the patient to enquire whether they have been completed and to answer any questions the patient may have.

ELIGIBILITY:
Inclusion Criteria:

* na

Exclusion Criteria:

* na

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Thomson, MBBS RANZCR, Principal Investigator — Bayside Health
Locations (1):
- Radiology Department, The Alfred, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Konstantatos AH, Kavnoudias H, Stegeman JR, Boyd D, Street M, Bailey M, Lyon SM, Thomson KR. A randomized, double-blind, placebo-controlled study of preemptive oral oxycodone with morphine patient-controlled anesthesia for postoperative pain management in patients undergoing uterine artery embolization for symptomatic uterine fibroids. Cardiovasc Intervent Radiol. 2014 Oct;37(5):1191-7. doi: 10.1007/s00270-014-0913-2. Epub 2014 Jul 1. PMID 24981461